CLINICAL TRIAL: NCT01899586
Title: Mechanisms and Functional Outcomes of Exercise Progression Models in the Elderly
Acronym: FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019806; 1RC1AG035822-01 (NIH)
Record Dates: First submitted 2013-07-11; First posted 2013-07-15 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Elderly; Sedentary
Keywords: Aging; Functional Capacity; Exercise Independence; Peripheral Adaptations; Vascular
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regional Specific Training (RSTS) (Experimental): The RSTS protocol was designed to focus on specific peripheral muscle groups without imposing a significant cardiorespiratory strain. Each exercise involved contractions with moderate load but with an extended duration of up to six minutes. Eight specific exercises were performed to target all major muscle groups and enable the routine to be completed within 60 minutes including warm-up, rest periods and stretching between exercises, and cool down exercises.
  Interventions: Other: Regional Specific Training Stimulus (RSTS)
- Aerobic Exercise (AE) (Experimental): Whole-body aerobic exercise at >50% of heart rate reserve (HRR) for 45 minutes, three days per week.
  Interventions: Other: Aerobic Exercise Regimen (AE)

INTERVENTIONS:
Other: Regional Specific Training Stimulus (RSTS) — The RSTS protocol was designed to focus on specific peripheral muscle groups without imposing a significant cardiorespiratory strain. Each exercise involved contractions with moderate load but with an extended duration of up to six minutes. Eight specific exercises were performed to target all major muscle groups and enable the routine to be completed within 60 minutes including warm-up, rest periods and stretching between exercises, and cool down exercises.
  Arms: Regional Specific Training (RSTS)
Other: Aerobic Exercise Regimen (AE) — Whole-body aerobic exercise at >50% of heart rate reserve (HRR) for 45 minutes, three days per week.
  Arms: Aerobic Exercise (AE)

SUMMARY:
The aim of this study is to devise a sufficiently high intensity training program that provided an optimal stimulus to remove the peripheral factors known to reduce functional capacity, and can be cardiovascular and orthopedically well tolerated by the elderly. Findings from study laboratories have suggested that a regional specific training stimulus (RSTS) results in rapid improvements in both vascular and muscular function. RSTS is a novel combination of resistance training and aerobic training applied simultaneously, and in a serial manner, to specific regions of the body. It involves high-intensity and frequency muscle contractions, generating a targeted exercise stimulus, without producing excessive cardiovascular or orthopedic stress. The hypothesis is that initiating training with RSTS at multiple, strategically selected peripheral sites, in a serial manner will elicit local vascular and muscular changes, thereby preparing individuals at elevated risk of losing independence, to respond and progress more favorably to whole-body exercise.

ELIGIBILITY:
Inclusion Criteria:

* >70 yrs of age
* Sedentary (exercising <1 day/wk)
* Non-smokers
* Able to ambulate without use of an assistive device
* Able to walk between 200-450m on a 6-minute walk test

Exclusion Criteria:

* Oxygen dependent
* Recent medications changes (within 3 months)
* Current Smokers
* Fixed-rate pacemakers
* Uncontrolled hypertension or Type II diabetes
* Positive ECG changes or angina during CPX testing
* Unable to complete a maximal CPX to volitional fatigue
* AHA Class D, or NYHA Class III or IV heart failure

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change In Exercise Capacity | Baseline, 4 weeks, and 12 weeks
  Exercise capacity was assessed using a maximal cardiopulmonary exercise (CPX) test with expired gas analysis, for determination of peak oxygen consumption and peak walking time.
Change in Maximal Strength | Baseline, 4 weeks, and 12 weeks
  Skeletal muscle strength was assessed using a one repetition maximum (1RM) measurement obtained for the seated row, chest press, leg press and handgrip.

SECONDARY OUTCOMES:
Change in Functional Ability | Baseline, 4 weeks and 12 Weeks
  The Senior Fitness Test is a previously validated battery of 6 physical tasks of daily living used to assess strength, flexibility and endurance in order to detect and predict future limitations in functional capacity. The test is designed to evaluate physical fitness domains including upper-body strength (Arm Curl), lower-body strength (Chair Sit-Stand), upper and lower body flexibility (Back Scratch and Chair Sit and Reach), balance and coordination (8 foot Up and Go), and endurance (Six Minute Walk).
Change In Vascular Function | Baseline, 4 weeks, and 12 weeks
  Ankle-brachial Index (ABI), Brachial artery flow-mediated dilation (BAFMD), and arterial stiffness (pulse wave velocity and pulse wave reflection).
Change in Skeletal Muscle Physiology | Baseline, 4 weeks, and 12 weeks
  Capillary density (mm2) and capillary to fiber ratio will be evaluated. Fiber type will be also determined to identify for types I, IIa and IIb muscle fibers.

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Allen, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Pennington Biomedical Center, Baton Rouge, Louisiana
  - Duke Center for Living; Wallace Clinic, Durham, North Carolina

REFERENCES:
- [Derived] Woessner MN, Welsch MA, VanBruggen MD, Johannsen NM, Credeur DP, Pieper CF, Sloane R, Earnest CP, Ortiz De Zevallos Munoz J, Church TS, Ravussin E, Kraus WE, Allen JD. Impact of a Novel Training Approach on Hemodynamic and Vascular Profiles in Older Adults. J Aging Phys Act. 2022 Apr 1;30(2):196-203. doi: 10.1123/japa.2020-0509. Epub 2021 Aug 4. PMID 34348230